CLINICAL TRIAL: NCT03446209
Title: Tocilizumab for the Treatment of Familial Mediterranean Fever - A Randomized, Doubleblind, Phase II Proof of Concept Study
Brief Title: Tocilizumab for the Treatment of Familial Mediterranean Fever
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TOFFIFE 1.1
Record Dates: First submitted 2017-12-11; First posted 2018-02-26 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2019-04

CONDITIONS: Familial Mediterranean Fever
MeSH Terms: conditions — Familial Mediterranean Fever | interventions — tocilizumab

STUDY DESIGN:
Intervention Model Description: Multi-center, phase II, randomized, placebo-controlled, double blind proof of concept trial
Who Masked: Participant, Investigator
Masking Description: Investigator and patient will be masked. There' ll be one qualified person in each center who s not going to be masked to prepare study treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tocilizumab (Experimental): Tocilizumab Infusion RoAcemtra (EU) or Actemra (Rest of the world)
  Interventions: Drug: Tocilizumab Infusion RoAcemtra (EU)
- Placebo (Placebo Comparator): 0,9% physiological Saline
  Interventions: Drug: Tocilizumab Infusion RoAcemtra (EU); Drug: 0.9% physiological saline

INTERVENTIONS:
Drug: Tocilizumab Infusion RoAcemtra (EU) — Experimental arm's patients will obtain TCZ intravenously once every 4 weeks for 28 weeks
  Other Names: Actemra
Drug: 0.9% physiological saline — Experimental arm's patients will obtain saline intravenously once every 4 weeks for 16 weeks. If necessary, patients will get "rescue medication" after week 16 to week 28.
  Arms: Placebo

SUMMARY:
Adult patients with Familial Mediterranean Fever, who have active disease

DETAILED DESCRIPTION:
FMF is a rare disease, which permanently affects daily life of the patients with severe pain and the risk of developing a life threatening amyloidosis. Today there are only very limited treatment options and an ongoing highly unmet medical need for improved treatment strategies. This study will be the first randomized, controlled trial to assess the benefit as well as the safety profile of IL6 receptor inhibition wirth TCZ in patients with FMF. Elevated tissue and serum levels of IL-6 have been implicated in the pathogenesis of FMF. FMF attacks are painfull during the period of the attack but are not life- or organthreatening and usually can be handeled by nonsteroidal and antipyretic treatment. Amyloidos is a longtime complication that appears after several years of uncontrolled disease. Placebo control trials' data are characterized as having greater ability to distinguish between effective and ineffective treatments (that is, greater assay sensitivity). The concerns about placebo use should revolve around the issue of risk to participants, rather than around denial of treatment, and that in the absence of a significant risk of harm, placebo treatment is acceptable. In general, it is easier to achieve statistical significance in placebo-controlled trials, where effects tend to be larger, such that smaller numbers of participants need to be exposed to the investigational medication (and research costs are lower.) This is especially important in rare diseases like FMF. If an active control was itself never evaluated in a placebo-controlled trial, using it in an equivalency study, begs the question of its efficacy. This is the case for Canakinumab as a potential active comparator in FMF. No randomized controlled trial is published for this indication by now. Therefore, a placebo controlled study over a period of 16 weeks seems to be justifiable without exposing our patients to risk of serious or irreversible harm. NSAR and antipyretic treatment, as a rescue therapy for attacks, is possible throughout the study. In addition, all patients with uncontrolled active disease despite NSAR or paracetamol will drop out and will be treated with escape therapy, especially Canakinumab. Based on the available safety data in the RA program, the adverse effects of TCZ have been shown to be manageable (e.g. cytopenia, liver encyme elevation), reversible and usually not treatment limiting . The safety profile and tolerability of TCZ are expected to be similar or even better in patients with FMF than in patients with rheumatoid arthritis or giant cell arteritis, as the cohort of FMF patients is, in general, younger and shows less concomitant diaseases. Overall, the benefit-risk ratio of FMF patients to be treated with TCZ is judged positive.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years and written informed consent
* FMF according to the Tel Hashomer Criteria; with at least one heterozygous or homozygous mutation of the MEFV gene
* Inadequate response or intolerance to colchicine (inadequate response/intolerance:

disease activity despite colchicine with at least 2 x 0.5 mg/day or intolerance to colchicine)

* Attack during the last 12 weeks, defined as episodes of fever and/or pericarditis and/or serositis and/or testis involvement and/or arthritis and/or erysipelas-like rash and

  * CRP > 0.5 mg/dl and/or ESR > 20mm/h and/or SAA > 10mg/dl
  * PGA >2
* Understand and voluntarily sign an informed consent document prior to any study related assessments/procedures.
* Ability to adhere to the study visit schedule and other protocol requirements.
* Females of childbearing potential (FCBP*) must agree to utilize two reliable forms of contraception simultaneously from heterosexual contact for at least 28 days before starting study drug, while participating in the study (including dose interruptions), and for 6 months after study treatment discontinuation and must agree to regular pregnancy testing during this timeframe to abstain from breastfeeding during study participation and 6 months after study drug discontinuation.
* Males must agree to use a latex condom during any sexual contact with FCBP while participating in the study and for 6 months following discontinuation from this study, even if he has undergone a successful vasectomy to refrain from donating semen or sperm while on Tocilizumab/Placebo and 6 months after discontinuation from this study treatment.
* All subjects must agree to refrain from donating blood while on study drug and 6 months after discontinuation from this study treatment.
* All subjects must agree not to share medication.

A female of childbearing potential is a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., who has had menses at any time in the preceding 24 consecutive months).

Exclusion Criteria:

Subjects presenting with any of the following criteria will not be included in the trial:

* Patient participating simultaneously in other clinical interventional trials
* Major surgery within 8 weeks prior to screening or planned major surgery within 12 months after randomization
* Transplanted organs (except corneal transplant performed more than 3 months prior to screening)

Exclusions Related to Prior or Concomitant Therapy

* Previous treatment with TCZ
* Treatment with glucocorticosteroids >10mg/day within 1 week; prednisolone ≤ 10mg/day can be given on a stable dose throughout the study
* Analgesic medication, other than paracetamol or ibuprofen or diclofenac or colchicine, which can be used at a stable dose throughout the study and/or for treatment of FMF attacks to the maximum allowed daily dose (paracetamol: 4000mg/day, ibuprofene: maximum 2400mg/day, diclofenac maximum 150mg/day; colchicine 12mg/day) .
* Treatment with any investigational agent within 12 weeks (or 5 half-lives of the investigational drug, whichever is longer) of screening
* Treatment with Anakinra within the last 1 week prior to baseline (ptb), Canakinumab within the last 8 week prior to baseline
* Treatment with etanercept within 2 weeks; certolizumab pegol, abatacept or adalimumab within 6 weeks; golimumab and infliximab within 8 weeks ptb
* Rituximab within 24 weeks ptb
* Leflunomide within 12 weeks ptb (washout possible),
* azathioprine, cyclophosphamide within 12 weeks ptb
* Immunization with a live/attenuated vaccine within ≤ 4 weeks ptb
* Previous treatment with cell-depleting therapies, including investigational agents or approved therapies: anti-CD33, anti-CD52, anti-CD4, anti-CD5, anti- CD3 and anti-CD19
* Treatment with intravenous gamma globulin within 6 months of baseline
* Treatment with plasmapheresis within 6 months of baseline
* Any previous treatment with alkylating agents such as chlorambucil, or with total lymphoid irradiation

Exclusions Related to General Safety

* History of severe allergic or anaphylactic reactions to human, humanized, or murine antibodies
* Evidence of serious uncontrolled concomitant cardiovascular, nervous system, pulmonary (including obstructive pulmonary disease), renal, hepatic, psychiatric or gastrointestinal (GI) disease
* History of diverticulitis, diverticulosis requiring antibiotic treatment, or chronic ulcerative lower GI disease such as Crohn's disease, ulcerative colitis, or other symptomatic lower GI conditions that might predispose a patient to perforations
* Known active current or history of recurrent bacterial, viral, fungal, mycobacterial, or other infections (including but not limited to tuberculosis (TB) and atypical mycobacterial disease, hepatitis B and C, and herpes zoster, but excluding fungal infections of the nail beds)
* Any major episode of infection requiring hospitalization or treatment with IV antibiotics within 4 weeks of screening or oral antibiotics within 2 weeks of screening
* Active TB requiring treatment within the previous 3 years; patients should be screened for latent TB and, if positive, treated according to local practice guidelines prior to initiating TCZ treatment; patients treated for TB with no recurrence within 3 years and patients treated for latent TB within 3 years are eligible.
* Primary or secondary immunodeficiency (history of or currently active)
* Evidence of malignant disease or malignancies diagnosed within the previous 5 years (except basal and squamous cell carcinoma of the skin or carcinoma in situ of the cervix uteri that have been excised and cured)
* FCBP who are not willing to use an effective method of contraception, such as condom, sterilization during the study and for a minimum of 6 months after study drug therapy and breast-feeding females
* Pregnant women
* Males of reproductive potential who are not willing to use an effective method of contraception, such as condom, sterilization, or true abstinence throughout study and for a minimum of 6 months after study drug therapy
* History of alcohol, drug, or chemical abuse within 1 year prior to screening

Laboratory Exclusions (at Screening)

* Serum creatinine >1.4 mg/dL in female patients and >1.6 mg/dL (in male patients
* ALT or AST > 2 ×ULN
* Total bilirubin > 2 x ULN
* Platelet count < 100 × 109/L
* Hemoglobin < 8.5 g/dL
* White blood cells < 3.0 ×109/L
* Absolute neutrophil count < 2.0 × 109/L
* Absolute lymphocyte count < 0.5 × 109/L
* Positive hepatitis B surface antigen, anti-HBc, HIV or hepatitis C antibody

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-04-23 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Efficacy: measured change of Physician's Global Assessment of disease activity (PGA) | at week -4,0,4,8,12,16,20,24,28,32
  Efficacy: measured by Physician's Global Assessment of disease activity (PGA) will be assessed at every visit
  The PGA will be based on a 5 point-scale (from 0 to 4):
  0=none (no) disease associated clinical signs and symptoms*
  1. minimal disease associated clinical signs and symptoms*
  2. mild disease associated clinical signs and symptoms*
  3. moderate disease associated clinical signs and symptoms*
  4. severe disease associated clinical signs and symptoms* *sign and symptoms for evaluation of PGA: chest pain, abdominal pain, arthralgia, arthritis, skin rash, fever (body temperature ≥ 38.0°C). Patient are asked to fill out a patient's diary to help the physician to judge the PGA primary endpoint will be the number of patients achieving an adequate response to treatment at week 16, defined as: PGA ≤ 2 + normalized ESR or CRP (the one that led to inclusion must be normalized) + normalized SAA

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events-Determination of Erytthro Sedimentation Rate (ESR) | at week -4,0,4,8,12,16,20,24,28,32
  To evaluate the safety of TCZ in subjects with FMF Safety of participating subjects will be assessed by regular clinical examinations, laboratory tests and reporting of adverse events. In case of a relapse the physician will discuss further treatment options with the patient and will initiate further treatment (according to local standard). Clinical laboratory testing for all study-relevant evaluations will be performed at all visits.
  Laboratory testing has to include:
  • ESR [mm after 1hour]
serological remission | at week 16, 28
  To evaluate the proportion of patients with the serological remission at week 16 + 28 (defined as CRP < 0.5 mg/dl)
SAA level | at week 16 + 28
  To evaluate the proportion of patients with normalized SAA level at week 16 + 28 (defined as SAA < 10mg/l)

OTHER OUTCOMES:
Incidence of Treatment-Emergent Adverse Events -Determination of the C-reactive protein | at week -4,0,4,8,12,16,20,24,28,32
  Safety of TCZ in subjects with FMF Safety of participating subjects will be assessed by regular clinical examinations, laboratory tests and reporting of adverse events. In case of a relapse the physician will discuss further treatment options with the patient and will initiate further treatment (according to local standard).
  CRP [mg/L]
Incidence of Treatment-Emergent Adverse Events -Determination of the blood cell count | at week -4,0,4,8,12,16,20,24,28,32
  Safety of TCZ in subjects with FMF Safety of participating subjects will be assessed by regular clinical examinations, laboratory tests and reporting of adverse events. In case of a relapse the physician will discuss further treatment options with the patient and will initiate further treatment (according to local standard).
  complete blood cell count with differential [cells/µl]
Incidence of Treatment-Emergent Adverse Events -Determination of serum parameters (Creatinine) | at week -4,0,4,8,12,16,20,24,28,32
  to evaluate the safety of TCZ in subjects with FMF Safety of participating subjects will be assessed by regular clinical examinations, laboratory tests and reporting of adverse events. In case of a relapse the physician will discuss further treatment options with the patient and will initiate further treatment (according to local standard).
  serum chemistry function tests :
  Creatinine [mg/dl]
Incidence of Treatment-Emergent Adverse Events -Determination of renal parameters (Uric Acid) | at week -4,0,4,8,12,16,20,24,28,32
  to evaluate the safety of TCZ in subjects with FMF Safety of participating subjects will be assessed by regular clinical examinations, laboratory tests and reporting of adverse events. In case of a relapse the physician will discuss further treatment options with the patient and will initiate further treatment (according to local standard).
  renal function tests :
  Uric Acid [mg/dl]
Incidence of Treatment-Emergent Adverse Events -Determination of serum and renal parameters (Glomerular Filtration Rate) | at week -4,0,4,8,12,16,20,24,28,32
  to evaluate the safety of TCZ in subjects with FMF Safety of participating subjects will be assessed by regular clinical examinations, laboratory tests and reporting of adverse events. In case of a relapse the physician will discuss further treatment options with the patient and will initiate further treatment (according to local standard).
  renal function tests :
  GFR [ml/min]
Incidence of Treatment-Emergent Adverse Events -Determination of liver parameters (Gamma Glutamyltransferase (GGT)) | at week -4,0,4,8,12,16,20,24,28,32
  Safety of TCZ in subjects with FMF Safety of participating subjects will be assessed by regular clinical examinations, laboratory tests and reporting of adverse events. In case of a relapse the physician will discuss further treatment options with the patient and will initiate further treatment (according to local standard).
  GGT[IU/L]
Incidence of Treatment-Emergent Adverse Events -Determination of liver parameters ( Alanine- (ALT) -Aminotransferase) | at week -4,0,4,8,12,16,20,24,28,32
  Safety of TCZ in subjects with FMF Safety of participating subjects will be assessed by regular clinical examinations, laboratory tests and reporting of adverse events. In case of a relapse the physician will discuss further treatment options with the patient and will initiate further treatment (according to local standard).
  ALT [IU/L]
Incidence of Treatment-Emergent Adverse Events -Determination of liver parameters ( Alanine-Aminotransferase (AST)) | at week -4,0,4,8,12,16,20,24,28,32
  Safety of TCZ in subjects with FMF Safety of participating subjects will be assessed by regular clinical examinations, laboratory tests and reporting of adverse events. In case of a relapse the physician will discuss further treatment options with the patient and will initiate further treatment (according to local standard).
  AST[IU/L]
Incidence of Treatment-Emergent Adverse Events -Determination of liver parameters (Biliribun) | at week -4,0,4,8,12,16,20,24,28,32
  to evaluate the safety of TCZ in subjects with FMF Safety of participating subjects will be assessed by regular clinical examinations, laboratory tests and reporting of adverse events. In case of a relapse the physician will discuss further treatment options with the patient and will initiate further treatment (according to local standard).
  Bilirubin [mg/dl]

CONTACTS AND LOCATIONS:
Locations (3):
- Germany (3):
  - Universitätsklinikum Köln, Klinik I für Innere Medizin, Cologne, North Rhine-Westphalia
  - Charité Universitätsmedizin Berlin, Klinik für Rheumatologie und Klinische Immunologie, Abteilung -Neue Therapien & Studien, Berlin
  - University Hospital Tuebingen; Department of oncology, hematology, rheumatology, immunology and pulmology, Tübingen

IPD SHARING:
Plan to Share IPD: No